CLINICAL TRIAL: NCT03559647
Title: The Effectiveness Of Atezolizumab Under Real-World Conditions In Patients With Locally-Advanced Or Metastatic Non-Small Cell Lung Cancer After Prior Chemotherapy
Brief Title: The Effectiveness Of Atezolizumab In Patients With Locally-Advanced Or Metastatic Non-Small Cell Lung Cancer After Prior Chemotherapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39885
Record Dates: First submitted 2018-05-07; First posted 2018-06-18 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants who have demonstrated a lack of Clinical Benefit from Atezolizumab
- Cohort 2: Participants who demonstrated durability of Clinical Benefit and Tumor Response to Atezolizumab
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered per the Summary of Product Characteristics (SmPC) from the European Medicines Agency (EMA).
  Groups: Cohort 2

SUMMARY:
Hyperion Is A Prospective, Multicenter, Non-Interventional, Two-Cohort Study Collecting Primary Data In Patients With Locally Advanced Or Metastatic NSCLC Of Squamous Or Non-Squamous Histology After Prior Chemotherapy Being Treated With Atezolizumab In Routine Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic NSCLC (histologically or cytologically confirmed stage IIIB/stage IV) and prior chemotherapy
* Decision to be treated with Atezolizumab according to Summary of Product Characteristics (SmPC) by treating physician, independent of this non-interventional study
* No contraindication to treatment with Atezolizumab

Retrospective Inclusion:

* Participants may be included retrospectively. Retrospective inclusion and documentation is limited to up to 9 weeks after initial start of therapy with Atezolizumab (corresponding to a maximum of 3 treatment cycles with drug administrations at 3-week intervals), corresponding to a maximum of 9 weeks prior to date of informed consent. Quality of life for this population will be captured and assessed retrospectively with a modified questionnaire for the period immediately prior to treatment start until study inclusion. participants who started Atezolizumab therapy more than 9 weeks prior to ICF being obtained may not be included in the study.
* Participants who give consent to be retrospectively enrolled but have already discontinued Atezolizumab for reasons such as loss of clinical benefit or toxicity may also take part in the study, given their first administration of Atezolizumab is within 9 weeks of consenting to take part, and they meet all other eligibility criteria.

Exclusion Criteria:

Patients not eligible for Atezolizumab treatment according to SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible are participants with locally advanced or metastatic NSCLC after prior chemotherapy, who have been chosen by their treating physicians to receive atezolizumab according to the current Summary of Product Characteristics (SmPC) of TECENTRIQ
Sampling Method: Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Time to loss of clinical benefit (TTLCB) from Atezolizumab treatment | Time from first dose to loss of clinical benefit as assessed by the treating physician, through the end of study (approximately 5 years).
Duration of response (DOR) to Atezolizumab treatment | Time from first documentation of complete response (CR) or partial response (PR), whichever occurs first, until progressive disease (PD), as evaluated by the physician according to routine practice or death; through the end of study (~ 5 years)

SECONDARY OUTCOMES:
Disease control rate (DCR) of overall population | Percentage of patients who achieved a CR, a PR, or stable disease (SD) as evaluated by the physician according to clinical practice at the time of the fifth Atezolizumab infusion; (until the end of study, approximately 5 years)
Progression-free survival (PFS) of overall population | Time from initiation of study treatment to the first occurrence of progressive disease (PD) or death from any cause, whichever occurs first, as evaluated by the physician according to clinical practice, through the end of study (approximately 5 years)
Time to response (TTR) of overall population | Time from first dose to first response as assessed in clinical routine, through the end of study (approximately 5 years)
Overall response rate (ORR) of overall population | Rate of CR and PR in patients as assessed in clinical routine, through end of study (approximately 5 years)
Best overall response (BOR) of overall population | Best response achieved within 12 weeks as assessed in clinical routine, through the end of study (approximately 5 years)
Best overall response of patients in cohort 2 ("Coh2 BOR") | Baseline through the end of study (approximately 5 years)
Overall survival of cohort 2 ("Coh2 OS") | Time from initiation of Atezolizumab treatment to death from any cause (until the end of study, approximately 5 years).
Percentage of participants with Adverse Events (AEs) | Baseline through the end of study (approximately 5 years)

OTHER OUTCOMES:
Health-related quality of life (HRQoL) | Prior to first Atezolizumab infusion, during Atezolizumab treatment, and post Atezolizumab discontinuation, through the end of study (approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (94):
- Germany (94):
  - Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Zentralklinikum Augsburg, Augsburg
  - Dres. Helmut Tanzer Joachim Hornberger und Johannes Kern, Bad Reichenhall
  - Klinikum Mittelbaden; Medizinisches Versorgungszentrum - Hämatologie und Onkologie, Baden-Baden
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Gynäkologie, Bamberg
  - St. Hedwig Kliniken Berlin GmbH, Berlin
  - Onkologisches Versorgungszentrum Friedrichshain; Hämatologie, Onkologie und Palliativmedizin, Berlin
  - Praxis Dr. Med. Gunhild Kühn, Berlin
  - Onkologie am Segelfliegerdamm, Berlin
  - Klinikum Bielefeld Mitte Klinik für Hämatologie, Onkologie u. Palliativmedizin, Bielefeld
  - Onkologische Schwerpunktpraxis Bielefeld; Haemotologie & Internistische onkologie, Bielefeld
  - Augusta Kranken-Anstalt gGmbH, Bochum
  - Klinikum Koeln-Merheim; Lungenklinik, Cologne
  - Fachkrankenhaus Coswig GmbH Zentrum f.Pneumologie Beatmungsmedizin Thorax-u.Gefäßchirurgie, Coswig
  - Med. Versorgungszentrum Filiale Donauwörth Onkologisches Zentrum, Donauwörth
  - Medizinische Klinik Nord, Lungenkrebszentrum, Dortmund
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Klinik St.Johannes-Hospital Medizinische Klinik I, Duisburg
  - Klinikum Barnim GmbH; Med. Klinik I, Gastroenterologie, Hämatologie, Onkologie, Eberswalde
  - Dres. Bruch, Buschmann, Linck, Euskirchen
  - Hämatologisch-Onkologische Fachpraxis Dr. med. Th. Ehlers & Dr. med. N. Karapanagiotidis, Frankenthal/Pfalz
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik I, Frankfurt
  - St. Elisabethen Krankenhaus, Frankfurt am Main
  - Klinikum Frankfurt Höchst GmbH; Klinik Innere Medizin 3 - Hämatologie, Onkologie, Palliativmedizin, Frankfurt am Main
  - Dres.Jochen Wilke und Harald Wagner, Fürth
  - Fachübergreifende Gemeinschaftspraxis Onkologie & Innere Medizin Dr. med. Haddadin & Panagiotou, Garbsen
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - SRH Wald-Klinikum Gera; Zentrum fur klinische Studien (ZKS), Gera
  - Agaplesion Pneumologische Klinik Waldhof Elgershausen; Pneumologie, Greifenstein
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Diakoniekrankenhaus Halle; Klinik für Pneumologie, Halle
  - Praxis für Hämatologie und Onkologie in Hamburg, Hamburg
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Hämatologische-Onkologische Schwerpunktpraxis, Hamburg
  - Dres.Andreas Karcher und Stefan Fuxius, Heidelberg
  - Onkologische Praxis in Heidenheim, Heidenheim
  - Onkologische Schwerpunktpraxis Hof; Dres. Hanns-Detlev; Harich und Christian Kasper, Hof
  - Klinikum Idar-Oberstein; Klinik für Neurochirurgie, Idar-Oberstein
  - Klinikum Konstanz; MVZ Onkologie, Konstanz
  - MVZ Hämatologie und Onkologie Krefeld, Krefeld
  - Internistische Praxis Hämatologie und Onkologie, Kronach
  - Klinikum Landshut Medizinische Klinik I, Landshut
  - Gemeinschaftspraxis für Hämatologie und Onkologie, PD Dr. Bauer, Dr. Thiel, Lebach
  - Dres. Barbara Tschechne Stefanie Luft und Wolf-Oliver Jordan, Lehrte
  - Universität Leipzig; Medizinische Klinik und Poliklinik I, Abteilung Pneumologie, Leipzig
  - ÜBAG MVZ Mitte / MVZ Delitzsch GmbH, Standort Leipzig, Leipzig
  - Bonifatius Hospital Lingen gGmbH; Hämatologie und Onkologie, Lingen
  - Lungenklinik Lostau, Lostau
  - Klinikum Ludwigsburg; Studiensekretariat, Ludwigsburg
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Klinikum Magdeburg gGmbH; Klinik für Hämatologie, Onkologie und Palliativmedizin, Magdeburg
  - Gemeinschaftspraxis Fr. Dr. med. Balser & Hr. Dr. med. Weidenbach, Marburg
  - Philipps-Universität Marburg; Klinik für Innere Med.; Schwerpunkt Hämatologie/Onkologie/Immunologie, Marburg
  - Praxis für Innere Medizin und Pneumologie, Markkleeberg
  - Dres. Michael Maasberg Marion Schmitz und Maria Theresia Keller, Mayen
  - Joh. Wesling Klinikum Minden; Klinik fuer Hämatologie und Onkologie, Minden
  - Gem.Praxis im Ärztezentrum Dr.med.Jörg Wiegand Jochen Eggert, Moers
  - Kliniken Ostalb, Stauferklinikum Schwäbisch-Gmünd; Zentrum für Innere Medizin, Mutlangen
  - Klinikum der Universität München; Medizinische Innenstadt, München
  - Lungenklinik Münnerstadt, Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Praxis Dr. Uhlig, Naunhof, Naunhof
  - Friedrich-Ebert-Krankenhaus Klinik f. Hämatologie/ Onkologie u. Nephrologie, Neumünster
  - Ruppiner Kliniken Medizinische Klinik A, Neuruppin
  - Praxis Dr. Losem, Neuss
  - Praxis für Hämatologie und Onkologie, Neuwied
  - Klinikum Nuernberg Nord; Medizinische Klinik 3, Pneumologie, Oncologie, Nuremberg
  - Pitri.Studien-GmbH (Ambulantes Therapiezentrum Hämatolgie/ Onkolgogie) Ärztehause 4 OG, Offenburg
  - Sana Kliniken Ostholtstein; Klinik Oldenburg; Innere Medizin; Onkologie, Oldenburg
  - Paracelsus-Klinik; Abteilung Haematologie und Onkologie, Osnabrück
  - Onkologische Studien GbR, Dres. Becker, Kreisel-Büstgens und Moorahrend, Porta Westfalica
  - Praxis für Hämatologie & Onkologie, Saarbrücken
  - Schwerpunktpraxis für Hämatologie und Onkologie Dr. Med. Thomas Edelmann, Schkeuditz
  - Zentrum Ambulante Onkologie, Schorndorf
  - Zentrum für ambulante Hämatologie und Onkologie; Onkologische Praxis, Siegburg
  - Onkologische Schwerpunktpraxis, Soest
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -; Klinik Dr. Hancken, Stade
  - Medizinisches Versorgungszentrum Stolberg, Stolberg
  - Praxisnetzwerk Hämatologie und InternistischeIOnkologie, Troisdorf
  - Universitätsklinikum Tübingen; Innere Medizin VIII, Medizinische Onkologie und Pneumologie, Tübingen
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - SHG-Kliniken Völklingen, Völklingen
  - Regio Klinikum Wedel; Pneumologie, Wedel
  - Praxis innere Medizin; Onkologie, Weimar
  - MedFISMO ltd., Weinsberg
  - Gemeinschaftspraxis für Hämatologie und Onkologie Westerstede Aurich Rhauder, Westerstede
  - Dres.Klaus Josten und Ortwin Klein, Wiesbaden
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven, Wilhelmshaven
  - Klinikverbund St. Antonius und St. Josef GmbH Petrus-Krankenhaus; Medi. Klinik III, Wuppertal
  - MVZ West GmbH Wuerselen; Haematologie-Onkologie, Würselen
  - Klinikum Würzburg Mitte gGmbH; Standort Missioklinik, Würzburg
  - Praxis Dr.med. Mathias Schulze, Zittau